CLINICAL TRIAL: NCT00516451
Title: Phase I Study of BMS-690514 in Japanese Patients With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA187-006
Record Dates: First submitted 2007-08-14; First posted 2007-08-15 (Estimated); Last update posted 2008-10-13 (Estimated); Status verified 2008-07

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — BMS-690514

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: BMS-690514

INTERVENTIONS:
Drug: BMS-690514 — Tablets, Oral, 100, 200, 250 or 300 mg once daily, 29 days or more

SUMMARY:
The purpose of this clinical study is to identify the maximum tolerated dose (MTD) of BMS-690514 once daily orally in Japanese subjects with advanced or metastatic solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with advanced or metastatic solid tumors for whom the standard of care is ineffective or inappropriate, with adequate kidney, liver and cardiac function.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2007-11; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
To determine the Maximum Tolerated Dose, the Dose Limiting Toxicity of BMS-690514 | administered orally every day 28 days

SECONDARY OUTCOMES:
Evaluate safety, exposure levels of BMS-690514 in the body & anticancer activity of BMS-690514 administered orally every day for 28 days. | throughout the study
Safety evaluations and laboratory assessments will be performed | throughout the study
Preliminary markers of efficacy will also be assessed | throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Chuo-Ku, Tokyo, Japan

REFERENCES:
- [Derived] Nokihara H, Yamamoto N, Yamada Y, Yamada K, Hirata T, Goto Y, Tanioka M, Ikeda Y, Tamura T. A phase I study of BMS-690514 in Japanese patients with advanced or metastatic solid tumors. Cancer Chemother Pharmacol. 2012 Oct;70(4):559-65. doi: 10.1007/s00280-012-1932-9. Epub 2012 Aug 10. PMID 22878519